CLINICAL TRIAL: NCT00303524
Title: An Open-label, Randomized, Parallel Group, Multicentre Study to Compare Oestradiol Suppression Between ZOLADEX 10.8 mg Depot Given 3 Monthly and ZOLADEX 3.6 mg Depot Given Monthly in Pre-menopausal Patients With ER Positive Early Breast Cancer
Brief Title: Comparative Study of Oestradiol Suppression: Zoladex 10.8mg/3 Month vs. 3.6mg/Month in ER +ve EBC Pre-menopausal Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8664C00004; Zoladex EBC Study
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

ARMS (2):
- 1 (Experimental): Zoladex 3-month depot
  Interventions: Drug: Goserelin acetate
- 2 (Experimental): Zoladex 1-month depot
  Interventions: Drug: Goserelin acetate

INTERVENTIONS:
Drug: Goserelin acetate — Injection 3.6 mg monthly
  Other Names: Zoladex
  Arms: 2
Drug: Goserelin acetate — injection 10.8 mg every 3 months
  Other Names: Zoladex
  Arms: 1

SUMMARY:
The primary purpose of this study is to establish if a 10.8 mg dose of ZOLADEX given 3 monthly is non-inferior to a 3.6 mg dose of ZOLADEX given monthly in terms of oestradiol suppression in patients with oestrogen receptor positive early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women aged 20 years or over with histological/cytologically-confirmed ER +ve breast cancer who have undergone radical surgery and WHO performance status 0,1 or 2.

Exclusion Criteria:

* Evidence of metastatic disease, previous bilateral oophorectomy or radiotherapy to the ovaries, previous chemotherapy, breast surgery completed over 12 weeks before starting trial treatment, previous neo-adjuvant/adjuvant hormonal breast cancer therapy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Zoladex 10.8mg depot (every 12 weeks) is non-inferior to Zoladex 3.6mg depot (every 4 weeks) in terms of oestradiol (E2) suppression in patient population by assessment of area under the curve of E2 concentration during the first 24 weeks of treatment. | every 12 weeks

SECONDARY OUTCOMES:
Zoladex 10.8mg has similar safety and tolerability profile to Zoladex 3.6mg. Examination of goserelin pharmacokinetics (PK) in Japanese patients after injection of Zoladex 10.8mg. Efficacy of Zoladex 10.8mg is similar to 3.6mg by assessment of DFS. | every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Japan Medical Director, MD, Study Director — AstraZeneca
Locations (22):
- Japan (22):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Isehara
  - Research Site, Kagoshima
  - Research Site, Kashiwa
  - Research Site, Kawasaki
  - Research Site, Kitakyushu
  - Research Site, Kumamoto
  - Research Site, Matsuyama
  - Research Site, Miyazaki
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ōta-ku
  - Research Site, Saitama
  - Research Site, Sayama
  - Research Site, Shimotsuke
  - Research Site, Suita
  - Research Site, Tokorozawa
  - Research Site, Tokyo
  - Research Site, Utsunomiya